CLINICAL TRIAL: NCT06771700
Title: Feasibility of an Intra-operative and Non-fluoroscopic Subcutaneous ICD Positioning and Assessment of the PRAETORIAN Score During Implantation: a Pilot Study
Brief Title: S-ICD Implantation: US Based Pilot Study
Acronym: SUSTAIN S-ICD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UKK2025_SICDImplant
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Sudden Cardiac Death
Keywords: S-ICD; Defibrillator
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Intervention Model Description: This is a pilot study. Patients are treated according to clinical standard. There are additional measurements made in the process but the study protocol does NOT include any deviation from the clinical standard practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S-ICD Implantation (Experimental): Patients are implanted with an S-ICD according to standard clinical practice. 1) The ideal lead and device position are determined using the new US method. Any deviation by more than 0.5 cm is counted as a significant deviation. 2) The intraoperative PRAETORIAN Score is calculated based on additional intraoperative measurements.
  Interventions: Diagnostic Test: Intraoperative PRAETORIAN Score

INTERVENTIONS:
Diagnostic Test: Intraoperative PRAETORIAN Score — The intraoperative PRAETORIAN Score is calculated based on the additional measurements.

SUMMARY:
This trial investigates two key aspects of the S-ICD implantation process. 1) For S-ICD implantation a pre-operative x-ray-based assessment of the anatomy and location of the heart is required. This study seeks to investigate the feasibility of US to potentially replace the need for x-ray 2) The PRAETORIAN score predicts defibrillation test success in subcutaneous ICD implantation but can only be calculated after the procedure. This pilot study aims to evaluate the feasibility of US determining the PRAETORIAN score intraoperatively. Lead-to-sternum distance and generator position measurments during the implantation procedure will be evaluated. Twenty consecutive patients scheduled for S-ICD implantation will be enrolled. The study involves no deviation from standard implantation procedures and requires no follow-up beyond standard post-operative chest X-ray on day one.

DETAILED DESCRIPTION:
This trial investigates two key aspects of S-ICD implantation. 1) To achieve successful shock conversion of an arrhythmia with the S-ICD, the optimal position of the electrode and the device are paramount. A pre-operative x-ray-based assessment of the anatomy and location of the heart is required. Using a dummy electrode and device placed on the patient's chest, the desired position is determined through fluoroscopy, and it is marked on the patient's skin. In this trial US will be used to determine the ideal lead and device position. As the current standard, the X-ray method will then confirm ideal positioning before the device is implanted.

2) The PRAETORIAN score is an established tool to predict defibrillation test success in subcutaneous ICD implantation but can only be calculated post-procedure using chest X-ray. This pilot study aims to evaluate the feasibility of determining the PRAETORIAN score intra-operatively. This pilot study will assess whether lead-to-sternum distance and generator position can be accurately measured during the implantation procedure by manual measurements with non-fluoroscopic means. This would potentially allow risk stratification before intra-operative defibrillation testing. Ten consecutive patients scheduled for S-ICD implantation will be enrolled. The study involves no deviation from standard implantation procedures and requires no follow-up beyond standard post-operative chest X-ray on day one. If successful, this approach could improve implantation safety by identifying high-risk patients before defibrillation testing.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients presenting for S-ICD implantation at our institution

Exclusion Criteria:

* patients unable to consent.
* pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
PRAETORIAN | 1 day after the device implantation, when chest x-ray is available
  The intraoperative PRAETORIAN Score is correlated with the regular PRAETORIAN Score

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - University Hospital Cologne, Cologne

IPD SHARING:
Plan to Share IPD: No
This is a pilot study with potential proprietary data